CLINICAL TRIAL: NCT00422136
Title: Genetic Epidemiology of Otitis Media
Brief Title: Genetics of Middle Ear Disease
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Margaretha L. Casselbrant, Principal Investigator, University of Pittsburgh
Other Study IDs: R01DC005630 (NIH); R01DC005630 (NIH)
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Otitis Media
Keywords: middle ear; otitis; genetics
MeSH Terms: conditions — Otitis Media; Otitis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples, DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to identify the genes that contribute to susceptibility to recurrent/persistent middle ear disease. Five hundred families with at least 2 children who have undergone tympanostomy tube insertion will be enrolled. A blood sample will be obtained from the children who had tubes and any available parent (at least 1), as well as any siblings without significant histories of middle ear disease.

DETAILED DESCRIPTION:
Using the twin study approach, the investigators demonstrated that time with middle ear effusion (MEE), number of episodes of MEE and numbers of episodes of acute otitis media (AOM) have a strong genetic component. The point estimate of heritability of time with MEE was 0.73. While there is significant evidence that susceptibility to recurrent/persistent OM is largely genetically determined, the specific genes which confer susceptibility are unknown. The overall research strategy to identify genes underlying OM is to apply a three-stage study design that will allow the investigators to balance cost efficiency with statistical power. Five hundred evaluable pairs of siblings with a history of tympanostomy tube insertion (affected), their parent(s) and available non-affected full siblings will be recruited. A blood sample will be obtained from each subject for genotyping.

ELIGIBILITY:
Inclusion Criteria:

* families: 2 or more full sibs who had tympanostomy tubes inserted

Exclusion Criteria:

* major congenital malformations
* medical conditions with a predisposition for OM (e.g. cleft palate, Down syndrome, or other craniofacial malformations
* cared for in the Intensive Care Unit as neonate
* been on assisted ventilation
* known sensorineural hearing loss

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Families with 2 or more full sibs who had tympanostomy tubes inserted
Sampling Method: Non-Probability Sample
Enrollment: 2121 (Actual)
Dates: Start 2002-07; Primary Completion 2007-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaretha L Casselbrant, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- ENT Research Center, Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Casselbrant ML, Mandel EM, Jung J, Ferrell RE, Tekely K, Szatkiewicz JP, Ray A, Weeks DE. Otitis media: a genome-wide linkage scan with evidence of susceptibility loci within the 17q12 and 10q22.3 regions. BMC Med Genet. 2009 Sep 3;10:85. doi: 10.1186/1471-2350-10-85. PMID 19728873